CLINICAL TRIAL: NCT00299975
Title: A Randomized Controlled Trial of Chinese Herbal Medicine in Three-dose Regimen for the Treatment of Functional Constipation
Brief Title: A Dose Determination Study of Chinese Herbal Medicine for Functional Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Professor, Director of Clinical Division, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID-001
Record Dates: First submitted 2006-03-06; First posted 2006-03-07 (Estimated); Results first posted 2011-12-16 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Constipation
Keywords: Randomized Controlled Trials; Medicine, Chinese Traditional; Medicine, Herbal; Constipation
MeSH Terms: conditions — Constipation | interventions — ma zi ren wan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MaZiRenWan (MZRW) Low dose (Experimental): MaZiRenWan (MZRW) Low dose 2.5g sachet by mouth, twice daily for 8 weeks
  Interventions: Drug: MaZiRenWan (MZRW) Low dose
- MaZiRenWan (MZRW) Median dose (Experimental): MaZiRenWan (MZRW) Median dose 5.0g sachet by mouth, twice daily for 8 weeks
  Interventions: Drug: MaZiRenWan (MZRW) Median dose
- MaZiRenWan (MZRW) High dose (Experimental): MaZiRenWan (MZRW) High dose 7.5g sachet by mouth, twice daily for 8 weeks
  Interventions: Drug: MaZiRenWan (MZRW) High dose

INTERVENTIONS:
Drug: MaZiRenWan (MZRW) Low dose — Dissolved MaZiRenWan (MZRW) granule (2.5g/sachet) in 150 ml hot water, take orally twice daily for 8 weeks
  Other Names: Hemp Seed Pill
  Arms: MaZiRenWan (MZRW) Low dose
Drug: MaZiRenWan (MZRW) Median dose — Dissolved MaZiRenWan (MZRW) granule (5.0g/sachet) in 150 ml hot water, take orally twice daily for 8 weeks
  Other Names: Hemp Seed Pill
  Arms: MaZiRenWan (MZRW) Median dose
Drug: MaZiRenWan (MZRW) High dose — Dissolved MaZiRenWan (MZRW) granule (7.5g/sachet) in 150 ml hot water, take orally twice daily for 8 weeks
  Other Names: Hemp Seed Pill
  Arms: MaZiRenWan (MZRW) High dose

SUMMARY:
Functional constipation (FC) is common with 14.3% estimated prevalence in Hong Kong, but treatment for this condition in conventional medicine is suboptimal. Complementary and alternative medicines, especially Chinese herbal medicine (CHM) are used frequently by patients with FC, but there is little research evidence about these commonly used CHM. The purpose of the study is evaluate the efficacy and safety of CHM, as well as determining the optimal dosage.

DETAILED DESCRIPTION:
Functional constipation (FC) is a common complaint in clinical practice, with the estimated prevalence 14.3% in Hong Kong, as nearly affecting 1 million Hong Kong People in different extent. It is comparable with western population, which is 15% in North America. By the definition of Rome II criteria, FC comprises a group of functional disorders, which presents as persistent difficult, infrequent or seemingly incomplete defecation.

Constipation is often perceived to be benign, easily treated condition with short-term treatment being relatively straightforward. However, the fact is the management of FC is perplexed as some subjects complain of constipation more than decade. Moreover, chronic constipation can develop into more serious bowel complaints, such as faecal impaction, incontinence and bowel perforations. There is also accumulating evidence shown that constipated subjects have significantly higher anxiety and depression scores and lower quality of life. Therefore, the demand of effective agents to normalize bowel function is extremely large.

Conventional treatment for constipation mainly relies on dietary fibre and laxatives. Although there is no credible evidence that any serious problem is associated with their prolonged use, the treatment of it has been suboptimal. First, a recent systematic review pointed out that there were paucity of trials for many commonly used agents, therefore, their use might not be well validated. Second, many patients with severe constipation do not respond adequately or lose of effectiveness after a short period of time. Third, many patients who intake dietary fibre complain of flatulence, distension, bloating and poor taste. As a result, the compliance is low as about 50%. Fourth, the use of osmotic laxatives, such as polyethylene glycol, become increasingly popular due to fewer side effects and better taste, however, the prices are much more expensive than other medications. Many constipation sufferers seek help from alternative medicine, especially from Chinese herbal medicine. For example, according to a telephone survey in Hong Kong, more than 85% of constipated subjects seek for coping strategies, such as asking for medical consultations, taking prescribed medicine and seeking for alternative therapy, involving Chinese medicine.

Traditional Chinese medicine (TCM) is particularly attractive as their effectiveness in treating functional disorders and retaining balance of body functions. The CHM used in study is derived from classic text of Chinese medicine (Shang Han Lun, Discussion of Cold-induced Disorders), which can "moisten the intestines, drain heat, promote the movement of qi and unblock the bowel".

It is well known that randomized controlled trial (RCT) is the gold standard to test the efficacy of intervention, thus in this project, we attempt to follow the basic requirements of RCT to testify the efficacy and safety of CHM on FC, as well as to determine the optimal dosage. We believe such study will benefit the advancement of CHM, or even as the foundation of research study in future.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of functional constipation with Rome II criteria
* General stool type belongs to Type 1 to 4 according to Bristol Stool Form Scale
* Complete spontaneous bowel movement≦2 movements per week

Exclusion Criteria:

* Anti-diarrhoeal therapy
* Drug-induced constipation
* Medical history of important bowel pathology, such as inflammatory bowel disease, congenital or acquired megacolon / megarectum
* Medical history of previous abdominal surgery
* Taking chronic medications that contain any kind of herbs, mineral, or specific vitamin supplements
* Medical history of carbohydrate malabsorption, hormonal disorder, cancer, diabetes mellitus, hypothyroidism, asthma, renal impairment and/or any other serious diseases
* History of laxative abuse
* History of allergy to Chinese herbal medicine
* Psychiatric or addictive disorders
* Pregnancy or breast-feeding
* Any other serious diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2006-10; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ZhaoXiang Bian, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Hong Kong Baptist University Chinese Medicine Clinic, Hong Kong, China

REFERENCES:
- [Result] Cheng CW, Bian ZX, Zhu LX, Wu JC, Sung JJ. Efficacy of a Chinese herbal proprietary medicine (Hemp Seed Pill) for functional constipation. Am J Gastroenterol. 2011 Jan;106(1):120-9. doi: 10.1038/ajg.2010.305. Epub 2010 Nov 2. PMID 21045817
- See also: Abstract — http://www.ncbi.nlm.nih.gov/pubmed/21045817

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All constipated patients (aged 18-65) who presented to the Chinese Medicine Clinics of School of Chinese Medicine, Hong Kong Baptist University from October 2006 to May 2007 were refered.
Pre-assignment Details: 177 patients were screened; of these 80 patients were excluded due to not meeting inclusion criteria (68 cases), refused to participate (6 cases) and lost to follow up (6 cases).
Groups:
- Low Dose Group: MaZiRenWan (MZRW) 2.5g/sachet Patients were instructed to dissolve a sachet of granules in 150 ml of hot water; they took this solution orally twice daily for 8 weeks.
- Median Dose Group: MaZiRenWan (MZRW) 5.0g/sachet Patients were instructed to dissolve a sachet of granules in 150 ml of hot water; they took this solution orally twice daily for 8 weeks.
- High Dose Group: MaZiRenWan (MZRW) 7.5g/sachet Patients were instructed to dissolve a sachet of granules in 150 ml of hot water; they took this solution orally twice daily for 8 weeks.
Period: Overall Study
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Started | 32 | 32 | 33
Received Allocated Intervention | 32 | 32 | 32
Completed | 29 | 31 | 25
Not Completed | 3 | 1 | 8
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group | Total
Number analyzed (Participants) | 32 | 32 | 32 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (9.8) | 38.8 (9.9) | 36.1 (9.2) | 36.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 30 | 87
  Male | 2 | 5 | 2 | 9
Duration of constipation [Mean (Standard Deviation); unit: years] | 10.9 (8.5) | 13.7 (10.0) | 15.0 (10.9) | 13.2 (9.9)
Bowel Movement [Mean (Standard Deviation); unit: movements per week] | 3.6 (1.5) | 3.1 (1.4) | 4.7 (4.1) | 3.8 (2.7)
Complete Spontaneous Bowel Movement (CSBM) [Mean (Standard Deviation); unit: movements per week] — CSBM referred to the feeling that defecation led to complete passage of stool rather than partial or incomplete evacuation without the use of any laxative or enema within 24 hours.
  movements per week | 0.5 (0.6) | 0.5 (0.7) | 0.5 (0.7) | 0.5 (0.7)
No. of days taking rescue therapy [Mean (Standard Deviation); unit: days per week] — Any medications, including laxatives, enemas and Chinese herbal medicine, for facilitating bowel movements.
  days per week | 1.7 (2.8) | 2.4 (3.3) | 2.2 (3.2) | 2.1 (3.1)
Severity of Constipation [Mean (Standard Deviation); unit: Units on a scale] — It was a 7-point ordinal scale from 0=not at all to 6=very severe.
  Units on a scale | 4.2 (1.1) | 4.1 (1.3) | 4.3 (1.5) | 4.2 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Responder for Complete Spontaneous Bowel Movement (CSBM)
Description: Participants with a mean increase of CSBM>=1 movement per week compared with the last 14 days of the run-in period were defined as responders.CSBM referred to the feeling that defecation led to complete passage of stool rather than partial or incomplete evacuation without the use of any laxative or enema within 24 hours.
Time Frame: Week3-10
Population: Statistical analysis was performed on the population being randomized and receiving allocated intervention. Missing values were imputed by the method of last observation carried forward.
Measure: Number; unit: participants
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Number analyzed (Participants) | 32 | 32 | 32
participants
  Responder | 10 | 14 | 17
  Non-responder | 22 | 18 | 15
Statistical Analysis 1: Comparison: Low Dose Group vs Median Dose Group vs High Dose Group; Test type: Superiority or Other; p < 0.05, Chi-squared; Chi-squared test from Crosstabs analysis

2. Secondary Outcome: Responder for Complete Spontaneous Bowel Movement (CSBM)
Description: Participants with a mean increase of CSBM>=1 movement per week compared with the last 14 days of the run-in period were defined as responders. CSBM referred to the feeling that defecation led to complete passage of stool rather than partial or incomplete evacuation without the use of any laxative or enema within 24 hours.
Time Frame: Week11-18
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Number analyzed (Participants) | 32 | 32 | 32
participants
  Responder | 9 | 10 | 11
  Non-responder | 23 | 22 | 21
Statistical Analysis 1: Comparison: Low Dose Group vs Median Dose Group vs High Dose Group; Test type: Superiority or Other; p < 0.05, Chi-squared; Chi-squared test from Crosstabs analysis

3. Secondary Outcome: Bowel Movement
Time Frame: Baseline(Week1-2), Within treatment(Week3-10) & Within follow-up(Week11-18)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: movements per week
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Number analyzed (Participants) | 32 | 32 | 32
movements per week
  Wk1-2 | 3.6 (1.5) | 3.1 (1.4) | 4.7 (4.1)
  Wk3-10 | 4.2 (1.7) | 4.8 (1.8) | 6.5 (5.5)
  Wk11-18 | 3.9 (1.6) | 3.5 (1.2) | 5.2 (4.2)
Statistical Analysis 1: Comparison: Low Dose Group vs Median Dose Group vs High Dose Group; Test type: Superiority or Other; p < 0.05, ANOVA

4. Secondary Outcome: Complete Spontaneous Bowel Movement (CSBM)
Description: CSBM referred to the feeling that defecation led to complete passage of stool rather than partial or incomplete evacuation without the use of any laxative or enema within 24 hours.
Time Frame: Baseline(Week1-2), Within treatment(Week3-10) & Within follow-up(Week11-18)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: movements per week
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Number analyzed (Participants) | 32 | 32 | 32
movements per week
  Week1-2 | 0.5 (0.6) | 0.5 (0.7) | 0.5 (0.7)
  Week3-10 | 1.4 (1.4) | 1.6 (1.5) | 2.0 (2.1)
  Week11-18 | 1.4 (1.5) | 1.0 (1.2) | 1.3 (1.6)
Statistical Analysis 1: Comparison: Low Dose Group vs Median Dose Group vs High Dose Group; Test type: Superiority or Other; p < 0.05, ANOVA

5. Secondary Outcome: Global Symptoms Improvement
Description: Participants were asked to rate their impression of change in constipation by comparing with their baseline (Wk2) at the visits during the treatment (Wk6), end of treatment (Wk10) and end of follow-up (Wk18) with scores from 0 to 6 represented markedly worse or better respectively. The response categories were collapsed to simply "improved" for score 4 to 6, "same" for score 3 or "worse" for score 0 to 2.
Time Frame: Week6, 10 & 18
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Number analyzed (Participants) | 32 | 32 | 32
participants
  Week6-Improved | 25 | 24 | 26
  Week6-Same | 4 | 7 | 4
  Week6-Worse | 3 | 1 | 2
  Week10-Improved | 20 | 27 | 24
  Week10-Same | 10 | 5 | 6
  Week10-Worse | 2 | 0 | 2
  Week18-Improved | 20 | 14 | 20
  Week18-Same | 11 | 14 | 12
  Week18-Worse | 1 | 4 | 0
Statistical Analysis 1: Comparison: Low Dose Group vs Median Dose Group vs High Dose Group; Test type: Superiority or Other; p < 0.05, Chi-squared; Chi-squared test from Crosstabs analysis was implemented between three treatment groups in each time frame

6. Secondary Outcome: Severity of Constipation
Description: It was a 7-point ordinal scale from 0=not at all to 6=very severe.
Time Frame: Baseline(Week2), Within treatment(Week6), End of treatment(Week10) & End of follow-up(Week18)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Number analyzed (Participants) | 32 | 32 | 32
Units on a scale
  Week2 | 4.22 (1.07) | 4.06 (1.32) | 4.25 (1.46)
  Week6 | 2.72 (1.87) | 2.03 (1.84) | 2.03 (1.75)
  Week10 | 2.62 (1.88) | 2.06 (1.76) | 2.06 (1.81)
  Week18 | 3.03 (1.91) | 2.91 (1.92) | 2.38 (1.74)
Statistical Analysis 1: Comparison: Low Dose Group vs Median Dose Group vs High Dose Group; Test type: Superiority or Other; p < 0.05, ANOVA

7. Secondary Outcome: Sensation of Straining
Description: It was a 7-point ordinal scale from 0=not at all to 6=very severe.
Time Frame: Baseline(Week2), Within treatment(Week6), End of treatment(Week10) & End of follow-up(Week18)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Number analyzed (Participants) | 32 | 32 | 32
Units on a scale
  Week2 | 4.03 (1.06) | 3.53 (1.61) | 3.78 (1.60)
  Week6 | 2.62 (1.79) | 1.84 (1.73) | 2.16 (1.61)
  Week10 | 2.56 (1.92) | 2.06 (1.70) | 1.94 (1.74)
  Week18 | 2.69 (1.86) | 2.78 (1.88) | 2.34 (1.60)
Statistical Analysis 1: Comparison: Low Dose Group vs Median Dose Group vs High Dose Group; Test type: Superiority or Other; p < 0.05, ANOVA

8. Secondary Outcome: Incomplete of Evacuation
Description: It was a 7-point ordinal scale from 0=not at all to 6=very severe.
Time Frame: Baseline(Week2), Within treatment(Week6), End of treatment(Week10) & End of follow-up(Week18)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Number analyzed (Participants) | 32 | 32 | 32
Units on a scale
  Week2 | 4.53 (1.41) | 3.5 (1.63) | 3.97 (1.26)
  Week6 | 2.81 (1.87) | 2.59 (1.66) | 2.59 (1.58)
  Week10 | 2.69 (1.91) | 2.63 (1.64) | 2.66 (1.77)
  Week18 | 3.00 (1.83) | 2.94 (1.70) | 2.50 (1.67)
Statistical Analysis 1: Comparison: Low Dose Group vs Median Dose Group vs High Dose Group; Test type: Superiority or Other; p < 0.05, ANOVA

9. Secondary Outcome: Sensation of Bloating
Description: It was a 7-point ordinal scale from 0=not at all to 6=very severe.
Time Frame: Baseline(Week2), Within treatment(Week6), End of treatment(Week10) & End of follow-up(Week18)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Number analyzed (Participants) | 32 | 32 | 32
Units on a scale
  Week2 | 2.53 (1.90) | 2.75 (1.92) | 3.28 (1.87)
  Week6 | 2.03 (1.91) | 1.84 (1.63) | 1.91 (1.82)
  Week10 | 1.78 (1.85) | 1.63 (1.66) | 1.75 (1.92)
  Week18 | 1.91 (1.69) | 2.19 (1.86) | 1.94 (1.76)
Statistical Analysis 1: Comparison: Low Dose Group vs Median Dose Group vs High Dose Group; Test type: Superiority or Other; p < 0.05, ANOVA

10. Secondary Outcome: Sensation of Abdominal Pain/Cramping
Description: It was a 7-point ordinal scale from 0=not at all to 6=very severe.
Time Frame: Baseline(Week2), Within treatment(Week6), End of treatment(Week10) & End of follow-up(Week18)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Number analyzed (Participants) | 32 | 32 | 32
Units on a scale
  Week2 | 1.00 (1.24) | 1.12 (1.29) | 1.59 (1.68)
  Week6 | 1.00 (1.27) | 1.03 (1.31) | 1.50 (1.48)
  Week10 | 0.41 (0.98) | 1.09 (1.20) | 1.47 (1.74)
  Week18 | 0.47 (0.92) | 0.91 (1.25) | 0.84 (1.19)
Statistical Analysis 1: Comparison: Low Dose Group vs Median Dose Group vs High Dose Group; Test type: Superiority or Other; p < 0.05, ANOVA

11. Secondary Outcome: Passing of Gas
Description: It was a 7-point ordinal scale from 0=not at all to 6=very severe.
Time Frame: Baseline(Week2), Within treatment(Week6), End of treatment(Week10) & End of follow-up(Week18)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Number analyzed (Participants) | 32 | 32 | 32
Units on a scale
  Week2 | 2.37 (1.70) | 2.59 (1.43) | 3.34 (1.29)
  Week6 | 2.03 (1.49) | 1.97 (1.49) | 2.44 (1.46)
  Week10 | 1.38 (1.24) | 2.06 (1.27) | 2.38 (1.56)
  Week18 | 1.25 (1.19) | 2.19 (1.36) | 2.53 (1.63)
Statistical Analysis 1: Comparison: Low Dose Group vs Median Dose Group vs High Dose Group; Test type: Superiority or Other; p < 0.05, ANOVA

12. Secondary Outcome: Adverse Effects (e.g. Renal and Liver Function Tests)
Time Frame: pre-treatment & post-treatment
Reporting Status: Not Posted
Measure: Mean (Standard Deviation)

13. Secondary Outcome: Blood Urea Level
Time Frame: Pre-treatment(Week2) & Post-treatment(Week10)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Number analyzed (Participants) | 32 | 32 | 32
mmol/L
  Week2 | 4.68 (1.23) | 4.54 (1.12) | 4.31 (1.25)
  Week10 | 4.40 (1.18) | 4.41 (0.94) | 4.30 (1.26)
Statistical Analysis 1: Comparison: Low Dose Group vs Median Dose Group vs High Dose Group; Test type: Superiority or Other; p < 0.05, Paired-Samples T Test; Paired-Samples T Test was implemented between pre-treatment (Wk2) and post-treatment (Wk10) of each treatment group

14. Secondary Outcome: Blood Creatinine Level
Time Frame: Pre-treatment(Week2) & Post-treatment(Week10)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Number analyzed (Participants) | 32 | 32 | 32
μmol/L
  Week2 | 58.81 (13.22) | 58.00 (15.23) | 57.38 (12.46)
  Week10 | 58.81 (10.17) | 60.06 (17.27) | 58.09 (13.74)
Statistical Analysis 1: Comparison: Low Dose Group vs Median Dose Group vs High Dose Group; Test type: Superiority or Other; p < 0.05, Paired-Samples T Test; Paired-Samples T Test was implemented between pre-treatment (Wk2) and post-treatment (Wk10) of each treatment group

15. Secondary Outcome: Serum Glutamic Pyruvic Transaminase(SGPT) Level
Time Frame: Pre-treatment(Week2) & Post-treatment(Week10)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Number analyzed (Participants) | 32 | 32 | 32
U/L
  Week2 | 32.38 (6.95) | 32.78 (5.33) | 34.06 (9.01)
  Week10 | 33.44 (8.99) | 34.06 (6.67) | 34.16 (7.32)
Statistical Analysis 1: Comparison: Low Dose Group vs Median Dose Group vs High Dose Group; Test type: Superiority or Other; p < 0.05, Paired-Samples T Test; Paired-Samples T Test was implemented between pre-treatment (Wk2) and post-treatment (Wk10) of each treatment group

16. Secondary Outcome: Serum Glutamic Oxaloacetic Transaminase(SGOT) Level
Time Frame: Pre-treatment(Week2) & Post-treatment(Week10)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Number analyzed (Participants) | 32 | 32 | 32
U/L
  Week2 | 18.50 (5.01) | 18.28 (4.30) | 19.44 (5.29)
  Week10 | 18.69 (5.04) | 19.09 (5.08) | 19.09 (5.57)
Statistical Analysis 1: Comparison: Low Dose Group vs Median Dose Group vs High Dose Group; Test type: Superiority or Other; p < 0.05, Paired-Samples T Test; Paired-Samples T Test was implemented between pre-treatment (Wk2) and post-treatment (Wk10) of each treatment group

ADVERSE EVENTS:
Time Frame: 18 weeks
Description: Within the whole study period
Arm/Group | Low Dose Group | Median Dose Group | High Dose Group
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 10/32 | 10/32 | 14/32
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Group (N=32) | Median Dose Group (N=32) | High Dose Group (N=32)
Abdominal pain/cramping or bloating (Gastrointestinal disorders) | 7 | 7 | 8
Upper gastro-intestinal discomfort (Gastrointestinal disorders) | 4 | 4 | 6
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 1
Disturbance of menstruation (Reproductive system and breast disorders) | 1 | 1 | 0
Puffy face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Increase body odor (General disorders) | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No